CLINICAL TRIAL: NCT04113733
Title: Combinatorial Single Cell Strategies for a Crohn's Disease Gut Cell Atlas
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Lori Coburn, Principle Investigator, Vanderbilt University Medical Center
Other Study IDs: 191738
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and colonic tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Crohn's Disease: This group consists of patients with a diagnosis of Crohn's disease undergoing colonoscopy for clinical care. Samples including tissue biopsy, blood and stool will be collected one time. In addition, patient information that may include questionnaires and medical record review will be collected.
  Interventions: Other: Sample Collection
- Control: This group will include patients undergoing screening colonoscopy as part of standard of care. Samples including tissue biopsy, blood and stool will be collected one time. In addition, patient information that may include questionnaires and medical record review will be collected.
  Interventions: Other: Sample Collection
- Cooperative Human Tissue Network: This group will consist of non-IBD patients and Crohn's disease patients participating in the Cooperative Human Tissue Network (CHTN). The CHTN will be utilized to obtain surgical specimens from these patients. The patients will be screened and consented via the CHTN protocol. No additional samples in the form of blood or stool will be collected. Associated clinical data will be collected through medical record review.

INTERVENTIONS:
Other: Sample Collection — Tissue biopsies will be performed at the time of colonoscopy along with blood and stool sample collection.
  Groups: Control; Crohn's Disease

SUMMARY:
Inflammatory bowel disease (IBD), consisting of two major forms, Crohn's disease (CD) and ulcerative colitis, affects more than 1.6 million people in the United States alone. Despite current therapies, remission only occurs in approximately half of patients. The goal of study is to map single-cell spatial relationships across the spectrum of ileum/ascending colon from healthy control patients to uninvolved/quiescent and involved/active CD patients and assess for relationships between single-cell data and patient clinical data.

The investigators will utilize endoscopic mucosal biopsies and surgical resection specimens with rapid transfer of fresh tissue to the single-cell preparation for RNA-sequencing and use of tissues for RNA-fluorescence in situ hybridization and multiplex immunofluorescence. Along with machine learning image analysis and bioinformatics, this will generate a robust/detailed single-cell gut cell atlas (GCA) of ileo-colonic CD at all disease activities versus normal tissues. The study will also compare the results of endoscopic mucosal biopsies to those obtained from full thickness surgical specimens by utilizing the Cooperative Human Tissue Network (CHTN).

The investigators anticipate the GCA data will provide new insights into disease pathogenesis, leading to new therapeutic targets.

ELIGIBILITY:
Inclusion criteria:

* Provision of consent form
* Male or female greater than or equal to 18 years old
* Healthy volunteers without IBD undergoing colonoscopy for colorectal cancer screening or patients with a diagnosis of Crohn's disease (CD) confirmed by endoscopy or radiology assessment undergoing colonoscopy for clinical care

Exclusion criteria:

* Pregnancy
* Coagulopathy or bleeding disorder
* Renal or hepatic impairment
* History of organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing standard of care colonoscopy procedure at Vanderbilt University Medical Center (VUMC) and/or receiving care at the VUMC Inflammatory Bowel Disease Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The change in cellular composition (i.e., percentage of cell types) between Crohn's disease and control patients as assessed by single-cell RNA sequencing analysis, RNA-fluorescence in situ hybridization, and multiplex immunofluorescence. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Coburn, MD, Principal Investigator — Vanderbilt University Medical Center; Keith T Wilson, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators agree to the timely release and sharing of information to be no later than the acceptance for publication of the main findings from the final data set. Investigators are also committed to ensuring that all data are free of identifiers that would permit linkage to individual research participants as well as variables that could lead to deductive disclosure of the identity of individual subjects.